CLINICAL TRIAL: NCT00970541
Title: Phase 1 Study That Will Compare 12 Weeks of Supplementation With Cinnamon Extract on the Action of Insulin and Blood Sugar (Glucose) With 12 Weeks of Supplementation With a Placebo.
Brief Title: Effect of Cinnamon Extract on Insulin Resistance in Polycystic Ovary Syndrome
Acronym: Eccentric
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Princiapal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 29010
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: Cinnamon; PCOS; low blood sugar; Insulin; Glucose
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Hypoglycemia | interventions — Flour

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinnamon Supplementation (Active Comparator): A 500mg (consumed as two, 250mg capsules) of cinnamon extract (Cinnamon Bark P.E> 20:1) will be consumed before meals, three times per day.
  Interventions: Dietary Supplement: Cinnamon Supplementation
- Placebo (Placebo Comparator): A 500 mg placebo (wheat flour) will be consumed before meals, three times per day.
  Interventions: Dietary Supplement: Placebo (wheat flour)

INTERVENTIONS:
Dietary Supplement: Cinnamon Supplementation — 1, 3, or 6g of cinnamon per day for 40 days
  Other Names: The bark of Cinnamoni Cassae
  Arms: Cinnamon Supplementation
Dietary Supplement: Placebo (wheat flour) — 1, 3, or 6g of placebo per day for 40 days
  Other Names: 500mg placebo (wheat flour) will be cnsumed before meals, three times per day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Cinnamon from the Cassae Plant is effective in the body as insulin could lower blood sugar levels.

DETAILED DESCRIPTION:
Insulin resistance is a condition in which body cells do not fully respond to the action of insulin, a hormone that controls the amount of sugar (glucose) in the blood. As a result, blood sugar levels become abnormally high. Insulin resistance is common in women with polycystic ovary syndrome (PCOS). This study involves the administration of a nutritional supplement (cinnamon extract). The cinnamon extract like regular cinnamon powder comes from the bark of Cinnamon Cassae plant. It is believed that cinnamon may act in the same way as insulin and therefore could potentially improve insulin resistance and help to lower blood sugar (glucose) levels.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years of age
* Have a body mass index 25-40 kg/m2
* Have a sedentary lifestyle (participated in less than 30 minutes of physical activity 3 days per week over the last 6 months)
* History of irregular menstrual cycles (fewer than 6 cycles in past year)
* Excess androgen (to be measured at screening)
* Willing to supplement normal diet with cinnamon extract and a placebo for 12 weeks
* You can stay overnight at Pennington Center three times over the next six months

Exclusion Criteria:

* Do not meet our diagnostic criteria for polycystic ovary syndrome
* Have heart disease, lung disease, liver disease, blood disease, kidney disease, type 1 or 2 diabetes, or any other disease that in the opinion of the doctor might make you ineligible.
* Have cancer (active malignancy with or without concurrent chemotherapy).
* Abuse alcohol or illegal drugs.
* Smoke or have smoked within the previous 6 months. No smoking will be permitted during the study.
* Have donated blood within 30 days prior to randomization date.
* Have a hemoglobin, hematocrit, red blood cell, or iron level below the normal lower limit at screening.
* Taking medications that alter your glucose metabolism, (30 minute or more, 4 or more times per week over the past year.)
* Unwilling or unable to adhere to the clinical evaluation schedule over the entire six-month follow-up period.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity measured by the euglycemic hyperinsulinemic clamp | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States